CLINICAL TRIAL: NCT06651190
Title: Building mHealth Parent Capacity to Manage Pain in Young Children With Cancer: A Pilot Randomized Controlled Trial
Brief Title: Pain Caregiver Resource (PainCaRe)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lindsay Jibb, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 1000081481
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will download the PainCaRe app from the web to their personal phone either virtually or in-person. Parents will receive app-based notifications to complete a pain assessment report once-daily. Assessments not completed will be marked as "missed". Parents will also have the ability to complete ad hoc pain assessments as needed.
  In response to the assessment indicating a child has pain, evidence-based, algorithm-driven pharmacological, physical, or psychological pain treatment guidance will be provided. This guidance is tailored to the age and developmental stage of the child.
  Interventions: Other: Pain Caregiver Resource (PainCaRe)
- Control Arm (No Intervention): Parents randomized to the control arm (non-intervention group) will not be assigned to the PainCaRe app and their child will continue to receive standard medical and pain care.

INTERVENTIONS:
Other: Pain Caregiver Resource (PainCaRe) — The purpose of the PainCaRe mobile health app is to support parents of young children with cancer (between the ages of 2-11 years) to manage their cancer-related pain at home. The app will ask caregivers to completed a brief 6-question pain assessment once daily and complete ad hoc assessments as needed. Based on the results of the pain assessment, real-time, evidence-based pain management suggestions, including will be provided to parents. The purpose of the pilot randomized controlled trial (RCT) is to evaluate the feasibility of implementing PainCaRe in a future RCT. Please find attached the study protocol for reference.
  Arms: Intervention Arm

SUMMARY:
Pain is a problem for children with cancer, especially when they are outside of the hospital setting. Younger children with cancer are particularly vulnerable to undermanaged pain because of their inability to self-report pain and their reliance on parents for treatment. One method to help these children to get the best care possible is through the use of smartphone-based mHealth solutions. Smartphone apps can provide treatment advice to patients experiencing pain in real-time and in any environment. This research will use a phased and user-centered approach with family caregivers to co-design and co-evaluate the new cancer Pain Caregiver Resource (PainCaRe) app to achieve the following aims: (1) high-fidelity software development and usability refinement; (2) evaluation of trial feasibility and preliminary effectiveness in a pilot randomized controlled trial (RCT); and (3) systematic analysis of caregiver app usage patterns to refine PainCaRe for optimal engagement prior to a future RCT.

ELIGIBILITY:
1. Be the primary caregiver, or person assuming the majority of care activities, for a child aged 2-11 years undergoing cancer treatment and experiencing above mild pain (≥3/10) in the week preceding study enrolment (pain measured by self or caregiver proxy using a validated numerical 11-point rating scale).
2. Be able to speak and read English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility - attrition | 1 year
  Percent of caregivers not completing 8-week outcome measures. Criteria for feasibility: attrition <25%.
Feasibility - accrual | 1 year
  Percent of eligible caregivers accrued per recruitment day. Criteria for feasibility: accrual >60%.
Feasibility - adherence | 8 weeks
  Adherence to the intervention will be measured using the Analytics Platform to Evaluate Effective Engagement (APEEE) platform, a proprietary analytics software measuring the number of once-daily pain assessments completed and engagement with pain treatment guidance. Criteria for feasibility: adherence to twice-daily pain reporting >65%.
Acceptability | 8 weeks
  Measured with the Acceptability E-Scale (AES). Criteria for acceptability: mean score of 4 on each item

SECONDARY OUTCOMES:
Child pain intensity - parent report | 8 weeks
  Measured by caregiver proxy report using the Brief Pain Inventory
Child pain intensity - child report | 8 weeks
  Measured by self-report for children ≥4 years of age using the Faces Pain Scale-Revised .
Child pain interference - parent report | 8 weeks
  Measured by parent proxy for children <8 years of age using appropriate version of PROMIS Pediatric Scale
Child pain interference - child report | 8 weeks
  Measured by self-report for children ≥8 years of age using appropriate version of PROMIS Pediatric Scale .
Child health-related quality of life - parent report | 8 weeks
  Measured by self-report for children <8 years of age using appropriate versions of the Pediatric Quality of Life Inventory 4.0 .
Child health-related quality of life - child report | 8 weeks
  Measured by self-report for children <8 years of age using appropriate versions of the Pediatric Quality of Life Inventory 4.0 .
Parent quality of life | 8 weeks
  Measured by parent report using the Caregiver Quality of Life Index - Cancer .
Parent pain management self-efficacy | 8 weeks
  Measured by parent report using the Pain Self-Efficacy Scale .
Parent care satisfaction | 8 weeks
  Measured by parent report using the Satisfaction with Child Healthcare Survey .

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will only be only be used as part of this study